CLINICAL TRIAL: NCT05747950
Title: The Effect of Local Vibration, Constraint-Induced Movement Therapy (CIMT) and Physiotherapy and Rehabilitation Applied to the Upper Extremity Spasticity and Decreased Functionality After Stroke
Brief Title: Different Treatment Methods Effect on Upper Extremity Spasticity and Decreased Functionality After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuhal Şevval Gökdere (Other)
Collaborators: Tokat State Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Zuhal Şevval Gökdere, physiotherapist, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.12.08
Record Dates: First submitted 2023-01-08; First posted 2023-02-28 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Spasticity as Sequela of Stroke; Limitation, Mobility
MeSH Terms: conditions — Stroke; Mobility Limitation | interventions — Vibration

STUDY DESIGN:
Intervention Model Description: In the study, 45 individuals between the ages of 18-75 who were diagnosed with stroke and met the inclusion criteria will be recruited. Individuals will be divided into 3 groups according to different treatment methods.
Who Masked: Participant, Investigator
Masking Description: Researcher: Kırıkkale University, Institute of Health Sciences, 2nd year graduate student with thesis, physiotherapist, Zuhal Şevval Gökdere Participants: In this study, Kırıkkale University Faculty of Medicine, Physical Therapy and Physical Therapy in Rehabilitation Hospital and Tokat State Hospital Volunteer treated in the unit, between 18-75 years old, diagnosed with stroke, 45 individual will be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vibration group (Other): Vibration is defined as "a mechanical stimulus characterized by oscillating movements".
  has been defined.The first method is a hand held as a local vibration application that can be applied directly to the widest part of the muscle with the object.is named. The second method, called whole body vibration, is a vibration source applied on the platform. Participants immediately after the sessions in addition to conventional physiotherapy.
  Upper extremity flexor on the hemiplegic side in supine position, 8 weeks, 3 sessions per week with a CE certified vibration device with a frequency of 50-110 Hz and an amplitude of 1-4 mm. Local vibration will be applied for 15 minutes each.
  Interventions: Other: Vibration
- Modified Constraint-Induced Movement Therapy group (Other): Modified Constraint-İnduced Movement Therapy is a rehabilitation technique that promotes 'repetitive' use of the affected upper extremity in people with upper extremity neurological motor deficits. Constraint-İnduced Movement Therapy upper extremity after stroke it is a rehabilitation approach used to increase functional use. post stroke Approximately 20-25% of surviving patients can meet the motor criteria of mCIMT. Participants In addition to conventional treatment, they can use their intact extremities at home with a shoulder stabilization orthosis.Restraint, grasping on the hemiplegic side, using spoons and forks, combing hair daily life activities, 8 weeks, 3 days a week, and approximately 3 hours Modified Constraint-İnduced Movement Therapy m(CIMT) will be applied.
  Interventions: Other: Modified Constraint-İnduced Movement Therapy
- Control group (Other): Control group in the training group, will be given a program that includes joint range of motion exercises, strengthening exercises, mobility and transfer activities, and various activities in order to increase participation in daily life activities as a routine conventional treatment in 60-minute sessions, 3 days a week, for 8 weeks.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Vibration — Vibration is used as an alternative to physical exercise in various areas to increase muscle performance and flexibility, improve balance and proprioception, reduce spasticity and increase bone density.
  Arms: Vibration group
Other: Modified Constraint-İnduced Movement Therapy — Compulsory use therapy is a form of treatment in which the movements of the healthy side are prevented and the use of the weak side is encouraged in the stroke patient.
  Arms: Modified Constraint-Induced Movement Therapy group
Other: Conventional Therapy — Conventional exercises
  Arms: Control group

SUMMARY:
The aim of our study is to objectively and clearly determine the differences between the Spasticity and Decreased Functionality in the Upper Extremity Flexor Group Muscles After Stroke, the Vibration, mBZHT and Physiotherapy and Rehabilitation Applications in terms of treatment process and effectiveness, and to increase the use of the hands and upper extremities in the daily life activities of the patient.

DETAILED DESCRIPTION:
The World Health Organization has defined stroke as a clinical condition that occurs suddenly, with no apparent cause other than a vascular cause, leading to focal or global cerebral dysfunction, lasting 24 hours or longer, or resulting in death. Stroke ranks third among the causes of death and first in terms of disability. Spasticity, a velocity-dependent increase in muscle tone as a part of upper motor neuron syndrome, is seen in a wide variety of neurological diseases, including stroke, and may occur in the first week after stroke.Rehabilitation aims to inhibit spasticity, improve motor functions, gain independence in activities of daily living, and improve health-related quality of life in stroke patients.This is an observational study within a study.This study was carried out in Kırıkkale University Faculty of Medicine, Physical Therapy and Rehabilitation Hospital and Tokat State Hospital Physical Therapy and Rehabilitation Unit 45 volunteers who were diagnosed with stroke, aged 18-75 years, who met the inclusion criteria of the study planned for the individual.In the study, patients were divided into 3 groups according to different treatment methods the effects of Local Vibration and m(CIMT) applied to upper extremity flexor muscle groups on spasticity and upper extremity functionality will be examined in addition to the conventional rehabilitation program in stroke individuals. A program that includes joint range of motion exercises, strengthening exercises, mobility and transfer activities and various activities to increase participation in daily life activities will be applied routinely for 3 sessions 45 minutes a week for 8 weeks in the first group of patients in the training group.In addition, in addition to conventional physiotherapy, patients in the 1st group immediately after the sessions. Upper extremity flexor on the hemiplegic side in supine position, 3 sessions per week with a CE certified vibration device with a frequency of 50-110 Hz and an amplitude of 1-4 mm.Vibration will be done for 15 minutes each.From the patients in the second group, for 8 weeks, 3 days a week, 60 minutes joint range of motion exercises as routine conventional treatment in sessions,strengthening exercises, mobility and transfer activities, and activities of daily living.In order to increase participation, a program including various activities will be implemented. Moreover after the sessions, patients can use their intact extremities with shoulder stabilization orthosis at home restraint, grasping on the hemiplegic side, using spoons and forks, combing hair daily life activities, 8 weeks, 3 days a week, and approximately 3 hours Modified Restrictor Forced Movement Therapy m(CIMT) will be applied.In the third group, the last group in the third group, for 8 weeks, 3 days a week, 60 minutes joint range of motion exercises as routine conventional treatment only in sessions, strengthening exercises, mobility and transfer activities, and activities of daily living. In order to increase participation, a program including various activities will be implemented.

First of all, all individuals; Demographic characteristics such as age, gender, height, weight, case report form will be questioned. Upper extremity of all subjects before and 8 weeks after treatment.

Spasticity (tonus, elasticity, stiffness) in flexor group muscles Modified Ashworth and It will be measured with modified Tardieu Scales. Manual dexterity, speed and coordination of upper extremity activities were determined by Fugl-Meyer Upper Limb Evaluation Scale, 9-Hole Peg Test, Box and Block Test [BBT]) and Upper Extremity Motor Activity Diary-28; The quality of life of individuals with stroke, with the Stroke-Specific Quality of Life Scale; Cognitive states of stroke individuals will be evaluated with the Mini Mental Test.

ELIGIBILITY:
Inclusion Criteria:

* Those who are diagnosed with stroke between the ages of 18-75 and can stand
* No cognitive and communication problems
* Persons weighing less than 150 kg
* Patients who have had at least 10 days after Botox application

Exclusion Criteria:

* Individuals who are not stable in terms of vital signs
* Those who have any open wounds on their upper extremities
* Those with spasticity and contracture that prevent sole contact
* Pathological conditions affecting upper extremity sensation (after surgery after fracture etc.)
* Those with a Mini Mental Test score below 24
* Posterior circulation stroke (stroke type in which basilar artery and cerebellum are affected)
* Arterial blood circulation disorders
* Lymphatic Edema
* Those who have been diagnosed with Multiple Sclerosis, Parkinson's and other neurological diseases
* People with vision and hearing problemsPatients who have been diagnosed with stroke for at least 8 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | Change in Upper Extremity Spasticity at 8 Weeks,Two measurements before and after treatment, 1 minute
  It is the most widely used clinical scale to evaluate spasticity. Despite its widespread clinical use, the reliability of the scale is questioned in some studies. Recent publications indicate that more studies are needed on the reliability of the scale.
Modified Tardieu Scale (MTS) | Change in Upper Extremity Spasticity at 8 Weeks,Two measurements before and after treatment, 1 minute
  Like the MAS, the Modified Tardieu Scale (MTS) is another clinical scale used to assess spasticity. Although it is not as widely used as MAS, it is recommended as a more effective method in the evaluation of spasticity because it measures resistance to passive movement at two different rates. While performing MTS, the extremities are moved passively with V1, V2 and V3 velocities. V1 speed; as slow as possible (slower than the gravity fall velocity of the limb segment), V2 velocity is defined as the extremity fall velocity, and V3 velocity is defined as as fast as possible (faster than the normal gravity fall velocity of the limb). In MTS, V1 velocity can be used to measure passive range of motion, and V2 or V3 velocities can be used to measure spasticity.

SECONDARY OUTCOMES:
Fugl-Meyer Upper Extremity Rating Scale | Change in Upper Extremity Functionality at 8 Weeks,Two measurements before and after treatment, 5 minutes
  It is a performance-based scale specific to hemiplegia, and each parameter is scored as 0: unsuccessful, 1: partially successful, 2: completely successful performance. Reflex activity, voluntary movements with dynamic flexor and/or extensor synergies, voluntary movements with the use of dynamic flexor and extensor synergies, voluntary movements without or little dependence on synergies, and normal reflex activity parameters are evaluated. When evaluating the wrist, three different functions of the wrist muscles are evaluated in the shoulder, elbow and forearm. In the hemiplegia hand evaluation, 7 movements (flexion, extension and five grip functions) are evaluated. In the evaluation of coordination / speed, finger-nose test is performed for the upper extremity. During this test, tremor, dysmetria, and speed of movement are evaluated. The maximum motor performance score for the upper extremity is 66 points.
Nine Hole Peg Test | Change in Upper Extremity Functionality at 8 Weeks,Two measurements before and after treatment, 4 minutes
  It is a simple, fast, manual skill test with proven validity and reliability. It is particularly sensitive to changes in upper extremity performance. The test material consists of nine small sticks made in standard sizes and a nine-hole board on which to place them. NHPT is applied with the patient in a sitting position. The patient is asked to line up the nine sticks in the box on the table as quickly as possible into the holes of the other box and, after finishing, remove them immediately. The test is started with the dominant hand, the time is measured with a stopwatch, and it is started when the hand touches the bars and ends when the last stick is placed in the box.
Stroke-Specific Quality of Life Scale | Change in Upper Extremity Functionality at 8 Weeks,Two measurements before and after treatment, 5 minutes
  In 1999, Williams et al. Developed by The original scale, consisting of 49 items in total, consists of 12 domains evaluating mobility, energy, upper extremity function, self-care, occupation/productivity, temperament, social role, family role, vision, language, thinking, and personality traits.
Box and Block Test (BBT) | Change in Upper Extremity Functionality at 8 Weeks,Two measurements before and after treatment, 1 minute
  The Box-Block Test was developed to assess rough manual dexterity and is a very simple, practical and quick test to use. A box and small wooden blocks are used for the test, which is divided into two equal areas right in the middle. Small wooden blocks are all placed on one side of the box. For the test, the patient is told to throw the wooden blocks in one section into the other section as quickly as possible and 60 seconds are given. The test is applied to both the dominant and non-dominant hand and the number of wooden blocks thrown to the opposite side gives the total score. The test is particularly suitable for patients with limited grip and dexterity.
Upper Extremity Motor Activity Diary-28 | Change in Upper Extremity Functionality at 8 Weeks,Two measurements before and after treatment, 5 minutes
  This scale, which aims to evaluate the function of the hemiparetic upper extremity, was developed by Uswatte et al. in 2006. 30 upper extremity functions are evaluated and scored with 2 different scales as "use level" and "use quality". The score for each scale is calculated by summing the scores and dividing by the number of marked items.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Kırıkkale, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Working Protocol with Other Researchers, Statistical Analysis Plan (SAP),Informed Consent Form (ICF),Clinical Trial Report (CSR) and Analytical Code will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 10, 2023 - June 10, 2023

REFERENCES:
- [Background] Nasb M, Li Z, S A Youssef A, Dayoub L, Chen H. Comparison of the effects of modified constraint-induced movement therapy and intensive conventional therapy with a botulinum-a toxin injection on upper limb motor function recovery in patients with stroke. Libyan J Med. 2019 Dec;14(1):1609304. doi: 10.1080/19932820.2019.1609304. PMID 31032717
- [Result] Caliandro P, Celletti C, Padua L, Minciotti I, Russo G, Granata G, La Torre G, Granieri E, Camerota F. Focal muscle vibration in the treatment of upper limb spasticity: a pilot randomized controlled trial in patients with chronic stroke. Arch Phys Med Rehabil. 2012 Sep;93(9):1656-61. doi: 10.1016/j.apmr.2012.04.002. Epub 2012 Apr 13. PMID 22507444
- [Result] Hsieh HC, Liao RD, Yang TH, Leong CP, Tso HH, Wu JY, Huang YC. The clinical effect of Kinesio taping and modified constraint-induced movement therapy on upper extremity function and spasticity in patients with stroke: a randomized controlled pilot study. Eur J Phys Rehabil Med. 2021 Aug;57(4):511-519. doi: 10.23736/S1973-9087.21.06542-4. Epub 2021 Jan 15. PMID 33448755